CLINICAL TRIAL: NCT02573311
Title: A 6-month OTC-simulated, Open Label, Uncontrolled Study of Tamsulosin 0.4 mg in Men
Brief Title: Actual Use Study of Tamsulosin in Men
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 527.85
Record Dates: First submitted 2015-10-01; First posted 2015-10-09 (Estimated); Results first posted 2020-04-08 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Urological Manifestations
MeSH Terms: conditions — Urological Manifestations | interventions — Tamsulosin

ARMS (1):
- men (Experimental)
  Interventions: Drug: tamsulosin hydrochloride

INTERVENTIONS:
Drug: tamsulosin hydrochloride

SUMMARY:
An actual use study to assess how men who respond to advertisements about urinary symptoms use tamsulosin in a simulated Over the Counter (OTC) setting including following "stop use and ask a doctor if" and "ask a doctor before use" statements and if they take the medication according to the label instructions, also assess any reported adverse events during simulated OTC use.

ELIGIBILITY:
Inclusion criteria:

* Men, 18 years of age and older, with bothersome urinary symptoms
* Able to speak, read and understand English
* Subject or anyone in their household is not currently employed by a marketing or marketing research company, advertising agency or public relations firm, a pharmacy or pharmaceutical company, a manufacturer of medicines, a managed care or health insurance company, as a certified or licensed healthcare professional or in a healthcare practice
* Has not participated in any clinical trial in the last 12 months
* Willing to sign an informed consent/HIPPA form and willing and able to provide contact information

Exclusion criteria:

* Allergy to tamsulosin hydrochloride or sulpha drugs
* Report current use of a medication listed on the "Do not use" section of the Drug Facts Label (DFL)
* Choose not to purchase the study product
* Do not provide consent or sign HIPPA form
* Do not provide contact information

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1117 (Actual)
Dates: Start 2015-09-23 (Actual); Primary Completion 2016-08-01 (Actual); Study Completion 2016-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (40):
- United States (40):
  - Parkway Discount Drugs, Birmingham, Alabama
  - Homewood Pharmacy, Homewood, Alabama
  - Robert's Discount Pharmacy, Hoover, Alabama
  - Pharmacy at the Pig, McCalla, Alabama
  - Pinson Discount Drugs, Pinson, Alabama
  - ACACIA Apothecary and Wellness, Tucson, Arizona
  - Parkview Compounding Pharmacy, Rancho Cucamonga, California
  - Garden Drug, Fort Lauderdale, Florida
  - Pill Box Pharmacy, Pembroke Pines, Florida
  - Sutton Family Pharmacy, Dalton, Georgia
  - Huff's Drug Store, Ellijay, Georgia
  - Wynn's Pharmacy Incorporated, Griffin, Georgia
  - Family Care Pharmacy, Highland, Illinois
  - Goodrich Pharmacy, Andover, Minnesota
  - Goodrich Pharmacy, Blaine, Minnesota
  - Goodrich Pharmacy, Elk River, Minnesota
  - Northfield Pharmacy, Northfield, Minnesota
  - Cub Pharmacy #1924, Saint Louis Park, Minnesota
  - The Medicine Shoppe and Elsberry Pharmacy, Elsberry, Missouri
  - Albers' Specialty Pharmacy, Kansas City, Missouri
  - Apex Specialty Pharmacy, Riverside, Missouri
  - Stevenson Family Pharmacy, Saint Joseph, Missouri
  - Countryside Pharmacy, Savannah, Missouri
  - Texas Road Pharmacy, Monroe, New Jersey
  - Duran Central Pharmacy, Albuquerque, New Mexico
  - Sam's Regent Pharmacy, Albuquerque, New Mexico
  - Total Care Pharmacy, Burlington, North Carolina
  - Kroger Pharmacy #342, Cary, North Carolina
  - Charleston Pharmacy, South Charleston, South Charleston, Ohio
  - Med Center Compounding Pharmacy & Health Center, Cleveland, Tennessee
  - T.B. Bond Pharmacy, Hillsboro, Texas
  - Eagle Pharmacy, Houston, Texas
  - Mountain West Apothecary, Bountiful, Utah
  - Maple Mountain Pharmacy, Mapleton, Utah
  - The Medicine Shoppe, Ogden, Utah
  - Family Plaza Pharmacy, West Jordan, Utah
  - Foothills Compounding Pharmacy, Enumclaw, Washington
  - Kelley-Ross Compounding Pharmacy, Seattle, Washington
  - Rxtra Care, Seattle, Washington
  - Kusler's Compounding Pharmacy, Snohomish, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The trial consisted of 2 parts. One was the product review phase (Part 1) and another was the actual use phase (Part 2). The number of enrolled patients in the protocol represent the number of participants (1117) who intended to purchase study product and enter part 2 of the study. All endpoints are based on part 2 of the study.
Groups:
- Cohort 1: Cohort 1 included all men who were not currently using a prescription medicine for Benign Prostatic Hyperplasia (BPH) and answered the purchase question for the study product (FLOMAX® (tamsulosin hydrochloride) 0.4 milligram (mg) capsules for self-directed use orally for a period of 24 weeks).
- Cohort 2: Cohort 2 included all men who were currently using a prescription medicine for Benign Prostatic Hyperplasia (BPH) and answered the purchase question for the study product (FLOMAX® (tamsulosin hydrochloride) 0.4 milligram (mg) capsules for self-directed use orally for a period of 24 weeks).
Period: Disposition for Part 1
Arm/Group | Cohort 1 | Cohort 2
Started | 1737 (Started are subjects who entered Part 1 and answered the purchase question) | 364 (Started are subjects who entered Part 1 and answered the purchase question)
Completed | 1730 (Completed are the subjects who actually completed Part 1) | 361 (Completed are the subjects who actually completed Part 1)
Not Completed | 7 | 3
Not completed — Withdrawal by Subject | 7 | 3
Period: Disposition for Part 2
Arm/Group | Cohort 1 | Cohort 2
Started | 964 (Started are subjects who purchased study product and are eligible to enter Part-2 of study.) | 153 (Started are subjects who purchased study product and are eligible to enter Part-2 of study.)
Completed | 754 (Completed are the subjects who completed use phase Part-2 (Week 24 and EOS-P2 interviews).) | 127 (Completed are the subjects who completed use phase Part-2 (Week 24 and EOS-P2 interviews).)
Not Completed | 210 | 26
Not completed — Physician Decision | 25 | 7
Not completed — Adverse Event | 36 | 5
Not completed — Lost to Follow-up | 76 | 7
Not completed — Withdrawal by Subject | 60 | 3
Not completed — Investigator decision | 0 | 1
Not completed — Other than specified above | 13 | 3

BASELINE CHARACTERISTICS:
Population: Analysis Set for Cohort 1 and 2: This set included all men who were currently not using a prescription medicine for BPH (Cohort 1) or were currently using a prescription medicine for BPH (Cohort 2) and who answered the purchase question in Part 1. (Age is missing for 8 men)
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 1731 | 362 | 2093
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.8 (11.67) | 68.3 (9.10) | 63.0 (11.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1731 | 362 | 2093

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Men Who Report a Condition Listed Under the "Stop Use and Ask a Doctor if" Section of the DFL Within the First 12 Weeks of Using Study Product and do Not Stop Use or Initiate Contact With Doctor Out of Total Population in Cohort 1
Description: Percentage of men who reported a condition listed under the "Stop use and ask a doctor if" section of the Drug Facts Label (DFL) within the first 12 weeks of using study product and did not stop use or initiated contact with a doctor out of the total population is presented along with 95% exact two sided Clopper-Pearson confidence interval.
Time Frame: 12 weeks
Population: Full Analysis Set for Actual Use (FAS-AU1) included all men who were currently not using a prescription medicine for BPH, purchased the study product, took at least one dose of study drug within the first 12 weeks of purchase and participated in at least 1 phone interview within the first 12 weeks of using the study product.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 924
Percentage of participants | 0.2 [0.0 to 0.8]

2. Secondary Outcome: Percentage of Men Who Report a Condition Listed Under the "Stop Use and Ask a Doctor if" Section of the DFL During the Study (24 Weeks) and do Not Stop Use or Initiate Contact With a Doctor Out of the Total Population in Cohort 1
Description: Percentage of men who reported a condition listed under the "Stop use and ask a doctor if" section of the DFL during the study (i.e., 24 weeks) and did not stop use or initiated contact with a doctor out of the total population of men in Cohort 1 is presented along with 95% exact two sided Clopper-Pearson confidence interval.
Time Frame: 24 weeks
Population: FAS AU1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 924
Percentage of participants | 0.2 [0.0 to 0.8]

3. Secondary Outcome: Percentage of Men Who Report Condition Listed Under "Stop Use and Ask a Doctor if" Section of the DFL and do Not Stop Use or Initiate Contact With Doctor Out of the Total Population in Cohort 1 Who Report the Condition Within 12 Weeks
Description: Percentage of men who reported a condition listed under the "Stop use and ask a doctor if" section of the DFL within 12 weeks of using study product and did not stop use or initiated contact with a doctor out of the total population of men in Cohort 1 who reported a condition listed under the "Stop use and ask a doctor if" section of the DFL within 12 weeks of using study product is presented along with 95% exact two sided Clopper-Pearson confidence interval.
Time Frame: Week 12
Population: Full Analysis Set for Actual Use and Stop Use and Ask If - Condition Within the First 12 Weeks: (FAS-AU1-COND12): These populations are subsets of the FAS-AU1 population which will include all men who report a condition listed under the "Stop use and ask a doctor if" section of DFL within the first 12 weeks of using the study product.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 207
Percentage of participants | 1.0 [0.1 to 3.4]

4. Secondary Outcome: Percentage of Men Who Report Condition Listed Under "Stop Use and Ask a Doctor if" Section of the DFL and do Not Stop Use or Initiate Contact With Doctor Out of the Total Population in Cohort 1 Who Report the Condition Within 24 Weeks
Description: Percentage of men who reported a condition listed under the "Stop use and ask a doctor if" section of the DFL within 24 weeks of using study product and did not stop use or initiated contact with a doctor out of the total population of men in Cohort 1 who reported a condition listed under the "Stop use and ask a doctor if" section of the DFL within 24 weeks of using study product is presented along with 95% exact two sided Clopper-Pearson confidence interval.
Time Frame: Week 24
Population: Full Analysis Set for Actual Use and Stop Use and Ask If - Condition Within the First 24 Weeks: (FAS-AU1-COND24): These populations are subsets of the FAS-AU1 population which will include all men who report a condition listed under the "Stop use and ask a doctor if" section of DFL within the first 24 weeks of using the study product.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 215
Percentage of participants | 0.9 [0.1 to 3.3]

5. Secondary Outcome: Percentage of Men Who Report a Condition Listed Under the "Stop Use and Ask a Doctor if" Section of the DFL Within the First 12 Weeks of Using Study Product Out of the Total Population in Cohort 1
Description: Percentage of men who reported a condition listed under the "Stop use and ask a doctor if" section of the DFL within the first 12 weeks of using the study product out of the total population of men in Cohort 1 is presented along with 95% exact two sided Clopper-Pearson confidence interval
Time Frame: 12 weeks
Population: FAS AU1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 924
Percentage of participants | 22.4 [19.8 to 25.2]

6. Secondary Outcome: Percentage of Men Who Report at Baseline a Symptom or Condition Under the "Ask A Doctor Before Use" Section of the DFL and Initiate Contact With a Doctor Out of the Total Population in Cohort 1
Description: Percentage of men who reported at baseline a symptom or condition under the "Ask A Doctor Before Use" section of the DFL and initiated contact with a doctor out of the total population of men in Cohort 1 is presented along with 95% exact two sided Clopper-Pearson confidence interval.
Time Frame: 24 weeks
Population: FAS AU1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 924
Percentage of participants | 20.3 [17.8 to 23.1]

7. Secondary Outcome: Percentage of Men Who Report at Baseline a Symptom or Condition Under the "Ask A Doctor Before Use" Section of the DFL and Initiate Contact With a Doctor Out of the Total Population of Cohort 1 Who Report a Symptom or Condition
Description: Percentage of men who reported at baseline a symptom or condition under the "Ask A Doctor Before Use" section of the DFL and initiated contact with a doctor out of the total population of men in Cohort 1 who reported a symptom or condition is presented along with 95% exact two sided Clopper-Pearson confidence interval.
Time Frame: 24 weeks
Population: Full Analysis Set for Actual Use and Ask a Doctor Before Use (FAS-AU1-ASK) is a subset of the FAS-AU1 population which included all men who reported a symptom or condition listed under the "Ask a doctor before use" section of the DFL.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 223
Percentage of participants | 84.3 [78.9 to 88.8]

8. Secondary Outcome: Percentage of Men Who Seek the Advice of a Physician Within the First 12/24 Weeks of the Study Out of the Total Population in Cohort 1
Description: Percentage of men who sought advice of a physician within the first 12/24 weeks of the study out of the total population of men in Cohort 1 is presented along with 95% exact two sided Clopper-Pearson confidence interval
Time Frame: Week 12 and Week 24
Population: FAS AU1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 924
Percentage of participants
  Week 12 (N=924) | 43.1 [39.9 to 46.3]
  Week 24 (N=924) | 56.4 [53.1 to 59.6]

9. Secondary Outcome: Percentage of Men Who Took Two or More Capsules Per Day Within the First 12/24 Weeks of Using Study Product Out of the Total Population in Cohort 1
Description: Percentage of men who took two or more capsules per day within the first 12/24 weeks of using study product out of the total population of men in Cohort 1 is presented along with 95% exact two sided Clopper-Pearson confidence interval
Time Frame: Week 12 and Week 24
Population: FAS AU1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 924
Percentage of participants
  Week 12 (N=924) | 7.6 [6.3 to 10.0]
  Week 24 (N=924) | 9.5 [8.1 to 12.1]

ADVERSE EVENTS:
Time Frame: From the first drug administration until 3 days after the treatment phase, up to 171 days.
Description: The Treated Set for Cohort (TS) included all men who were currently not using a prescription medicine for BPH (TS1) or were currently using a prescription medicine for BPH (TS2), purchased the study product and took at least one dose of study drug.
Groups:
- Cohort 1: Cohort 1 included all men who were not currently using a prescription medicine for Benign Prostatic Hyperplasia (BPH) and answered the purchase question for the study product (FLOMAX® (tamsulosin hydrochloride) 0.4 milligram (mg) capsules for self-directed use orally for a period of 24 weeks). (TS1)
- Cohort 2: Cohort 2 included all men who were currently using a prescription medicine for Benign Prostatic Hyperplasia (BPH) and answered the purchase question for the study product (FLOMAX® (tamsulosin hydrochloride) 0.4 milligram (mg) capsules for self-directed use orally for a period of 24 weeks). (TS2)
- Cohort 1 and 2: Cohort 1 and 2 included all men who answered the purchase question for the study product (FLOMAX® (tamsulosin hydrochloride) 0.4 milligram (mg) capsules for self-directed use orally for a period of 24 weeks) regardless of whether they were currently using the product or not. (TS)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 1 and 2
Serious Adverse Events (participants affected / at risk) | 54/927 | 12/150 | 66/1077
Other Adverse Events (participants affected / at risk) | 61/927 | 25/150 | 86/1077
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=927) | Cohort 2 (N=150) | Cohort 1 and 2 (N=1077)
Atrial flutter (Cardiac disorders) | 1 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 1
Cardiovascular disorder (Cardiac disorders) | 1 | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 1 | 2
Coronary artery occlusion (Cardiac disorders) | 1 | 1 | 2
Myocardial infarction (Cardiac disorders) | 2 | 1 | 3
Glaucoma (Eye disorders) | 1 | 0 | 1
Retinal detachment (Eye disorders) | 1 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1
Chest pain (General disorders) | 2 | 1 | 3
Hypersensitivity (Immune system disorders) | 0 | 1 | 1
Anal abscess (Infections and infestations) | 1 | 0 | 1
Appendicitis perforated (Infections and infestations) | 1 | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 1
Influenza (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 2
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Sepsis (Infections and infestations) | 1 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 3
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Carotid artery disease (Nervous system disorders) | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 1
Seizure (Nervous system disorders) | 1 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 1
Calculus urinary (Renal and urinary disorders) | 1 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Hospitalisation (Surgical and medical procedures) | 2 | 0 | 2
Aortic aneurysm (Vascular disorders) | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 1
Hypertension (Vascular disorders) | 2 | 0 | 2
Hypotension (Vascular disorders) | 1 | 1 | 2
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=927) | Cohort 2 (N=150) | Cohort 1 and 2 (N=1077)
Nasopharyngitis (Infections and infestations) | 48 | 17 | 65
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 8 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.